CLINICAL TRIAL: NCT03362320
Title: A Randomized Clinical Trial Comparing Arthroscopic Double- Versus Single-layer Reconstruction of the Rotator Cuff: Clinical and Radiological Outcome
Brief Title: Arthroscopic Rotator Cuff Tear Repair: Single Versus Double Layer Fixation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Austrian Research Group for Regenerative and Orthopedic Medicine (Other)
Responsible Party: Principal Investigator, Philipp Heuberer, Principal Investigator, Austrian Research Group for Regenerative and Orthopedic Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLvsDL
Record Dates: First submitted 2017-11-16; First posted 2017-12-05 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- double layer fixation (Experimental): Patients with torn infraspinatus and supraspinatus tendon undergoing arthroscopy rotator cuff repair with double layer fixation
  Interventions: Procedure: double layer fixation
- single layer fixation (Experimental): Patients with torn infraspinatus and supraspinatus tendon undergoing arthroscopy rotator cuff repair with single layer fixation
  Interventions: Procedure: single layer fixation

INTERVENTIONS:
Procedure: double layer fixation
  Arms: double layer fixation
Procedure: single layer fixation
  Arms: single layer fixation

SUMMARY:
Retear rates after arthroscopic rotator cuff repairs remain unsatisfactorily high. Recently, attention has been paid to restore the rotator cuff's native anatomy by reconstructing the superior joint capsule. However, the debate whether to reconstruct only the superficial tendinous part or also the deeper capsulo-ligamentous part of the rotator cuff is ongoing. Thus, the intention of the present study is to compare double-layer versus single-layer arthroscopic rotator cuff repair regarding retear rate and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients with repairable supra- and infraspinatus tears scheduled for arthroscopic rotator cuff fixation
* tear size of at least 2.5 cm and up to 4.0 cm
* signed informed consent

Exclusion Criteria:

* axillary nerve palsy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Retear rate | 12 months postoperatively
  Comparison of re-ruptures rate evaluated with magnetic resonance imaging between groups

SECONDARY OUTCOMES:
Constant-Murley score | baseline, 24 and 60 months postoperatively
  Comparison of the total Constant-Murley score (min 0 to max 100; higher values represent a better outcome) between groups
Range of motion (ROM) | baseline, 24 and 60 months postoperatively
  Comparison of ROMs between groups
Satisfaction with the procedure | 24 and 60 months postoperatively
  Comparison of satisfaction with the procedure between groups. Satisfaction is evaluated by asking patients one question to rate their satisfaction with the procedure based on a likert scale (4 = 'very satisfied', 3 = 'quite satisfied', 2 = 'moderately satisfied', 1 = 'less satisfied', 0 = 'not at all satisfied').
VAS | baseline, 24 and 60 months postoperatively
  Comparison of the Visual Analogue Scale (VAS) between groups
SST | baseline and 24 months postoperatively
  Comparison of the Simple Shoulder Test (SST) between groups
ASES | baseline, 24 and 60 months postoperatively
  Comparison of the American Shoulder and Elbow Surgeons score (ASES) between groups. The ASES is a patient-rated questionnaire with a total between 0 and 100 points with higher scores indicating better outcome.
qDASH | baseline, 24 and 60 months postoperatively
  Comparison of the quick Disability of the Arm, Shoulder and Hand (qDASH) between groups
WORC | baseline and 24 months postoperatively
  Comparison of the Western Ontario Rotator Cuff Index (WORC) between groups
SSV | baseline, 24 and 60 months postoperatively
  Comparison of the Simple Soulder Value (SSV) between groups
SF-36 | baseline, 24 and 60 months postoperatively
  Comparison of the quality-of-life score short form 36 (SF-36) between groups
Tendon integrity | baseline and 60 months postoperatively
  Comparison of tendon integrity (re-tear / no re-tear) evaluated with magnetic resonance imaging between groups

CONTACTS AND LOCATIONS:
Overall Officials: Werner Anderl, MD, Study Director — Austrian Research Group for Regenerative and Orthopedic Medicine; Philipp R Heuberer, MD, Principal Investigator — Austrian Research Group for Regenerative and Orthopedic Medicine
Locations (1):
- St. Vincent Shoulder & Sports Clinic, Vienna, Austria

REFERENCES:
- [Derived] Heuberer PR, Pauzenberger L, Gruber MS, Ostermann RC, Hexel M, Laky B, Anderl W. Delaminated Rotator Cuff Tears Showed Lower Short-term Retear Rates After Arthroscopic Double-Layer Repair Versus Bursal Layer-Only Repair: A Randomized Controlled Trial. Am J Sports Med. 2020 Mar;48(3):689-696. doi: 10.1177/0363546519897033. Epub 2020 Jan 9. PMID 31917608